CLINICAL TRIAL: NCT02229812
Title: Safe Implementation of Thrombolysis in Stroke - Monitoring Study (SITS-MOST)
Brief Title: Safe Implementation of Thrombolysis in Stroke - Monitoring Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 135.313
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- thrombolytic therapy in stroke
  Interventions: Drug: alteplase

INTERVENTIONS:
Drug: alteplase

SUMMARY:
Study to evaluate the safety and efficacy of intravenous alteplase within 3 hours of symptom onset in acute ischemic stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Female or male in-patient
* Age 18 - 80 years
* Clinical diagnosis of ischemic stroke causing a measurable neurological deficit defined as impairment of language, motor function, cognition, gaze, vision and/or neglect. Ischemic stroke is defined as an event characterized by sudden onset of acute focal neurological deficit, presumed to be caused by cerebral ischemia, after CT scan exclusion of hemorrhage
* Onset of symptoms within 3 hours prior to initiation of thrombolysis treatment
* Stroke symptoms present for at least 30 minutes that had not significantly improved before treatment. Symptoms must be distinguishable from an episode of generalized ischemia (i.e. syncope), seizure, or migraine disorder
* Patients are willing to receive thrombolysis treatment and to give informed consent with regard to retrieval of data and follow up procedures, according to the regulations in participating countries
* Willingness and ability to comply with the study protocol

Exclusion Criteria:

* Evidence of intracranial hemorrhage (ICH) on the CT-scan
* Symptoms of ischemic attack began more than 3 hours prior to infusion start or when time of symptom onset is unknown
* Minor neurological deficit or symptoms rapidly improving before start of infusion
* Severe stroke as assessed clinically and/or by appropriate imaging techniques
* Seizure at onset of stroke
* Symptoms suggestive of subarachnoid hemorrhage, even if the CT-scan is normal
* Administration of heparin within the previous 48 hours and a thromboplastin time exceeding the upper limit of normal for laboratory
* Patients with any history of prior stroke and concomitant diabetes
* Prior stroke within the last 3 months
* Platelet count of below 100,000/mm³
* Systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, or aggressive management (IV medication) necessary to reduce BP to these limits
* Blood glucose <50 or > 400 mg/dl
* Known hemorrhagic diathesis
* Patients receiving oral anticoagulants, e.g. warfarin sodium
* Manifest or recent severe or dangerous bleeding
* Known history of or suspected intracranial hemorrhage
* Suspected subarachnoid hemorrhage or condition after subarachnoid hemorrhage from aneurysm
* Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)
* Hemorrhagic retinopathy, e.g. in diabetes (vision disturbances may indicate hemorrhagic retinopathy)
* Recent (less than 10 days) traumatic external heart massage, obstetrical delivery, recent puncture of a non-compressible blood-vessel (e.g. subclavian or jugular vein puncture
* Bacterial endocarditis, pericarditis
* Acute pancreatitis
* Documented ulcerative gastrointestinal disease during the last 3 months, oesophageal varices, arterial- aneurysm, arterial/venous malformation
* Neoplasm with increased bleeding risk
* Severe liver disease, including hepatic failure, cirrhosis, portal hypertension oesophageal varices) and active hepatitis
* Major surgery or significant trauma in past 3 months

All in- and exclusion criteria follow the summary of product characteristics of Actilyse®

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute stroke patients in the European Union
Sampling Method: Non-Probability Sample
Enrollment: 6475 (Actual)
Dates: Start 2002-12; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of symptomatic intracerebral hemorrhage (SICH) | up to 36 hours
Mortality rate | 3 months

SECONDARY OUTCOMES:
Independence for activities of daily living | 3 months
  modified Ranking Scale 0-2